CLINICAL TRIAL: NCT04156971
Title: Effects of Omega-3 Long-Chain Polyunsaturated Fatty Acids (N-3 LCPUFA) Supplementation on Body Composition, Biochemical Profile, Diet and Physical Activity of Obese Children
Brief Title: Effects of Omega-3 Supplementation on Nutritional Status and Physical Activity of Obese Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Putra Malaysia (Other)
Responsible Party: Principal Investigator, Nor Baizura Md. Yusop, Senior Lecturer, Universiti Putra Malaysia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: JPD_Feb(13)05(Interview)
Record Dates: First submitted 2019-10-30; First posted 2019-11-08 (Actual); Last update posted 2019-11-13 (Actual); Status verified 2019-11

CONDITIONS: Life Style Modification; Childhood Obesity
Keywords: Childhood obesity; Life style modification; Omega 3; supplementation
MeSH Terms: conditions — Pediatric Obesity | interventions — Docosahexaenoic Acids

STUDY DESIGN:
Intervention Model Description: A parallel study is a type of clinical study where two groups of treatments. The intervention group (IG) received stage-based lifestyle modification intervention and fish oil supplement, while the control group (CG) received stage-based lifestyle modification intervention only.
Who Masked: Participant, Care Provider
Masking Description: After the parents/caregivers completed the consent form, the participants were age matched and randomized using a permuted block method, with a block size of four, into either IG or CG. To guarantee allocation concealment, we had the recommendation the randomization carried out by an independent third party.
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention Group (Experimental): stage-based lifestyle modification intervention and fish oil supplement (omega-3). Stage-based Lifestyle Modification consists of several activities that include nutrition counselling, aerobic sessions, a hands-on activity 'Let's Play' and 'Sharing is Caring' Participants in the intervention group were also given fish oil capsules containing n-3 LCPUFA (DHA and EPA) for a duration of 16 weeks. The participants were required to consume two fish oil capsules, providing 1320 mg n-3 LCPUFA (792 mg EPA, 20:5n-3 and 528 mg DHA, 22:6n-3), and 6 IU vitamin E (D-alpha tocopherol) daily. The EPA and DHA ratio was 1.5:1.
  Interventions: Dietary Supplement: Omega 3; Behavioral: stage-based lifestyle modification intervention
- Control Group (Other): Only received Stage-based Lifestyle Modification consists of several activities that include nutrition counselling, aerobic sessions, a hands-on activity 'Let's Play' and 'Sharing is Caring'
  Interventions: Behavioral: stage-based lifestyle modification intervention

INTERVENTIONS:
Dietary Supplement: Omega 3
  Arms: Intervention Group
Behavioral: stage-based lifestyle modification intervention

SUMMARY:
Omega-3 Long-Chain Polyunsaturated Fatty Acids has potential as a supplement that can accelerate the effects of a weight management program in children. This study assessed the effects of fish oil supplementation on biochemical profile, body composition, diet and physical activity of obese children. A total of 37 obese children (7-11 years) were randomized to intervention (n=19) or control (n=18) group. Data were collected at baseline, at follow-up (every four weeks) and at 24 of the interventions. The intervention group (IG) received stage-based lifestyle modification intervention and fish oil supplement, while the control group (CG) received stage-based lifestyle modification intervention only. Changes in biochemical profile, body composition, diet and physical activity were examined in both intervention and control groups.

DETAILED DESCRIPTION:
Main objective To determine the effect of stage-based lifestyle modification and n-3 LCPUFA (DHA and EPA) supplements on body composition, biochemical profile, diet and physical activity of obese children.

Specific objectives

1. To compare changes in: i. Primary outcome: BMI-for-age ii. Secondary outcomes: Body composition (waist circumference [WC], mid-upper arm muscle circumference [MUAMC] and body fat percentage)

Biochemical profile:

Lipid profile (total cholesterol [TC], triglyceride [TG], low-density lipoprotein [LDL] and high-density lipoprotein [HDL]), fasting blood glucose (FBG), insulin and Homeostasis model assessment insulin-resistance index (HOMA-IR index), Fatty acid composition (DHA and EPA) Others: Adiponectin, high-sensitivity C-reactive protein (hs-CRP) and serum ferritin iii. Energy and nutrient intakes (Macronutrients, Saturated Fatty Acids [SFA], Polyunsaturated Fatty Acids [PUFA], Monounsaturated Fatty Acids [MUFA], Cholesterol and sugar and dietary fiber) vii. Physical activity between children receiving Stage-based Lifestyle Modification for the Management of Childhood Obesity with or without supplementation of 1320 mg of n-3 LCPUFA (DHA and EPA).

Intervention Group

Participants in the intervention group received Stage-based Lifestyle Modification and 16 weeks' supplementation of n-3 LCPUFA (DHA and EPA).

1. Stage-based Lifestyle Modification

   Stage-based Lifestyle Modification consists of several activities that include nutrition counselling, aerobic sessions, a hands-on activity 'Let's Play' and 'Sharing is Caring'. The recommendation for the dietary and physical activity modification was based on the NPG for the Management of Childhood Obesity (developed in Phase I). During the nutrition counselling session, educational topics related to dietary (reduce intake of fat and increase intake of fruits and vegetables) and physical activity modification (reduce sedentary activity and increase physical activity) were delivered based on the TTM.

   Participants' SOC for dietary and physical activity were determined before any information was given. This was important to ensure that the selected educational topic was tailored to the participant's current SOC. For each counselling session, at least two goals, one for dietary and one for physical activity, were set. Parents/caregivers were encouraged to participate in the nutrition counselling session. An aerobic session was conducted to encourage participants to be more active and increase their motivation levels, while a hands-on activity 'Let's Play' was aimed at increasing the knowledge of participants about food choices, food selection and healthy food preparation. The last activity was the 'Sharing is Caring' session to encourage parents/caregivers to share their experiences during the intervention period.
2. Supplementation of n-3 LCPUFA (DHA and EPA)

Participants in the intervention group were given fish oil capsules containing n-3 LCPUFA (DHA and EPA) for a duration of 16 weeks. The participants were required to consume two fish oil capsules, providing 1320 mg n-3 LCPUFA (792 mg EPA, 20:5n-3 and 528 mg DHA, 22:6n-3), and 6 IU vitamin E (D-alpha tocopherol) daily. The EPA and DHA ratio were, 1.5:1. The role of vitamin E is to stabilise the oil and is equal to 57%, 53.6% and 42.6% of Vitamin E RNI for Malaysia (2005) for children aged 7 to 9 years old, 10 to 12-year-old girls and 10 to 12-year-old boys, respectively. Participants were instructed to consume the capsules once a day before breakfast.

Determination of Dosage

Prior to supplementation with n-3 LCPUFA (DHA and EPA), other guidelines and outcomes of previous studies were reviewed. The recommendation of n-3 LCPUFA intake is 0.3 to 1.2% of total calorie intake. Supplementation of 0.6% of DHA/EPA from total energy is an acceptable range and an effective dosage for weight reduction in children and below the potential level that could lead to complications

The required dosage for the study ranged from 1186.7 mg to 1326.6 mg per day. Thus, the participants were asked to consume two fish oil capsules per day, which is equal to 1320 mg/day. Girls aged 7 to 9 years in the study consumed about 260 mg of DHA and EPA above their suggested amount. However, the amount is still below the potential level that could lead to complications. Each participant received sufficient fish oil capsules (60 capsules) for one month (30 days) of the intervention period.

Control Group Participants received Stage-based Lifestyle Modification for the management of childhood obesity only.

Study Measurements Information on demographic and socioeconomic, medical status, Child Feeding Questionnaire (CFQ), Family Eating and Activity Habits Questionnaire (FEAHQ) and Nutrition Knowledge at baseline were obtained though face-to-face interviews between researcher and parents/caregivers. With the help of their parents/caregivers, participants completed the Physical Activity Questionnaire for Older Children (PAQ-C) and three-day food record. Clear instructions were given to the parents/caregivers before they answered the questionnaires. In each visit, participants' anthropometric measurements were obtained and their BP was taken. Blood analysis was conducted at baseline, week 16 and week 24 for lipid profile, FBG, insulin and HOMA-IR index, fatty acid composition (DHA and EPA), adiponectin, hs-CRP and serum ferritin.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 7 to 11 years old.
* Classified as obese (>+2SD) based on BMI-for-age for 5 to 19 years old (WHO, 2007).

Exclusion Criteria:

• Children diagnosed with asthma, diabetes mellitus (DM), psychiatric disorders (e.g.

schizophrenia, severe autism or mental retardation, or psychosis), or other serious medical conditions.

* Children receiving medications that could potentially promote weight gain or weight loss.was sent to lab for lipid profile, FBG, insulin, hs-CRP and ferritin analysis.
* Children participating in any weight management programmes.
* Overweight, normal weight and underweight children.

Ages: 7 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 37 (Actual)
Dates: Start 2013-06-01 (Actual); Primary Completion 2014-07-31 (Actual); Study Completion 2015-02-28 (Actual)

PRIMARY OUTCOMES:
BMI-for-age change | Change from Baseline SBMI-for-age at 24 weeks
  Height and weight were measured to calculate BMI-for-age

SECONDARY OUTCOMES:
waist circumference [cm] | Every four weeks for a duration of 24 weeks
  Participants with abdominal obesity were determined based on the 90th percentile values for WC for sex and age
Mid-Upper Arm Muscle Circumference [cm] Mid-Upper Arm Muscle Circumference | Every four weeks for a duration of 24 weeks
  A fibreglass tape (measuring tape SECA 201 SECA Vogel and Halke Gmbh & Co., Germany) was used to measure MAC at non-vascular access sites of participants. Participants were required to stand in an erect position with the upper arm approximately parallel to the body and their forearms placed palm down across the middle of the body with the elbow bent to 90 degrees. The midpoint of the tip of the acromion process and the olecranon process was marked. The middle of the arm perpendicular to the long axis of the divisional was measured using a fibreglass tape. The measurement was recorded to the nearest 0.1 cm. The following formula was used to calculate MUAMC.
  Mid-Upper Arm Muscle Circumference
Total cholesterol [TC] mmol/L | week 0, week 16 and week 24
  A trained nurse and lab assistant performed blood drawing in the Haematology Lab, Faculty of Medicine and Health Sciences, Universiti Putra Malaysia. Five ml blood samples were collected three times; baseline, week 16 and week 24. All participants were required to fast overnight (10 to 12 hours), except for one to two glasses of plain water before the blood draw session. A fasting blood sample was collected from a peripheral vein of the arm for lipid profile, FBG, insulin, hs-CRP and ferritin analysis.
Triglyceride mmol/L | week 0, week 16 and week 24
  A trained nurse and lab assistant performed blood drawing in the Haematology Lab, Faculty of Medicine and Health Sciences, Universiti Putra Malaysia. Five ml blood samples were collected three times; baseline, week 16 and week 24. All participants were required to fast overnight (10 to 12 hours), except for one to two glasses of plain water before the blood draw session. A fasting blood sample was collected from a peripheral vein of the arm for lipid profile, FBG, insulin, hs-CRP and ferritin analysis.
Low-density lipoprotein [LDL] mmol/L | week 0, week 16 and week 24
  A trained nurse and lab assistant performed blood drawing in the Haematology Lab, Faculty of Medicine and Health Sciences, Universiti Putra Malaysia. Five ml blood samples were collected three times; baseline, week 16 and week 24. All participants were required to fast overnight (10 to 12 hours), except for one to two glasses of plain water before the blood draw session. A fasting blood sample was collected from a peripheral vein of the arm for lipid profile, FBG, insulin, hs-CRP and ferritin analysis.
High-density lipoprotein [HDL]) mmol/L | week 0, week 16 and week 24
  Fasting blood glucose (FBG), insulin and homeostasis model assessment insulin-A trained nurse and lab assistant performed blood drawing in the Haematology Lab, Faculty of Medicine and Health Sciences, Universiti Putra Malaysia. Five ml blood samples were collected three times; baseline, week 16 and week 24. All participants were required to fast overnight (10 to 12 hours), except for one to two glasses of plain water before the blood draw session. A fasting blood sample was collected from a peripheral vein of the arm for lipid profile, FBG, insulin, hs-CRP and ferritin analysis.
Fasting blood glucose (FBG) mmol/L | week 0, week 16 and week 24
  A trained nurse and lab assistant performed blood drawing in the Haematology Lab, Faculty of Medicine and Health Sciences, Universiti Putra Malaysia. Five ml blood samples were collected three times; baseline, week 16 and week 24. All participants were required to fast overnight (10 to 12 hours), except for one to two glasses of plain water before the blood draw session. A fasting blood sample was collected from a peripheral vein of the arm for lipid profile, FBG, insulin, hs-CRP and ferritin analysis.
Insulin [uU/mL] | week 0, week 16 and week 24
  A trained nurse and lab assistant performed blood drawing in the Haematology Lab, Faculty of Medicine and Health Sciences, Universiti Putra Malaysia. Five ml blood samples were collected three times; baseline, week 16 and week 24. All participants were required to fast overnight (10 to 12 hours), except for one to two glasses of plain water before the blood draw session. A fasting blood sample was collected from a peripheral vein of the arm for lipid profile, FBG, insulin, hs-CRP and ferritin analysis.
Homeostasis model assessment insulin-resistance index (HOMA-IR index) | week 0, week 16 and week 24
  HOMA-IR index, as a measure of insulin resistance, was calculated as [fasting insulin (μU/mL)]X[fasting glucose (mmol/L)]/22.5
DHA | week 0, week 16 and week 24
  Plasma lipid extraction process was carried out based on the principle of the Folch Method. For analysis of fatty acids' on the same day with the preparation of FAME, a total of 500 μl of hexane was added to the FAME and it was dried and analysed using gas chromatography (GC) 6890N (Network GC System).
EPA | week 0, week 16 and week 24
  Plasma lipid extraction process was carried out based on the principle of the Folch Method. For analysis of fatty acids' on the same day with the preparation of FAME, a total of 500 μl of hexane was added to the FAME and it was dried and analysed using gas chromatography (GC) 6890N (Network GC System).
Adiponectin | week 0, week 16 and week 24
  Plasma levels of adiponectin were determined using a novel enzyme-linked immunosorbent assay (ELISA) (ALPCO Diagnostics, Salem, NH) (ADIPOA).
High-sensitivity C-reactive protein (hs-CRP)[mg/L] | week 0, week 16 and week 24
  A trained nurse and lab assistant performed blood drawing in the Haematology Lab, Faculty of Medicine and Health Sciences, Universiti Putra Malaysia. Five ml blood samples were collected three times; baseline, week 16 and week 24. All participants were required to fast overnight (10 to 12 hours), except for one to two glasses of plain water before the blood draw session. A fasting blood sample was collected from a peripheral vein of the arm for lipid profile, FBG, insulin, hs-CRP and ferritin analysis.
Serum ferritin[ng/mL] | week 0, week 16 and week 24
  A trained nurse and lab assistant performed blood drawing in the Haematology Lab, Faculty of Medicine and Health Sciences, Universiti Putra Malaysia. Five ml blood samples were collected three times; baseline, week 16 and week 24. All participants were required to fast overnight (10 to 12 hours), except for one to two glasses of plain water before the blood draw session. A fasting blood sample was collected from a peripheral vein of the arm for lipid profile, FBG, insulin, hs-CRP and ferritin analysis.
calorie | Every four weeks for a duration of 24 weeks
  Three day food record
Carbohydrate [g & %] | Every four weeks for a duration of 24 weeks
  Three day food record
Protein [g & %] | Every four weeks for a duration of 24 weeks
  Three day food record
Fat [g & %] | Every four weeks for a duration of 24 weeks
  Three day food record
Saturated fatty acid [g & %] | Every four weeks for a duration of 24 weeks
  Three day food record
Polyunsaturated fatty acid [g & %] | Every four weeks for a duration of 24 weeks
  Three day food record
monounsaturated fatty acid [g & %] | Every four weeks for a duration of 24 weeks
  Three day food record
Fibre [g & %] | Every four weeks for a duration of 24 weeks
  Three day food record
Sugar [g & %] | Every four weeks for a duration of 24 weeks
  Three day food record
Physical activity level | Every four weeks for a duration of 24 weeks
  Physical Activity Questionnaire for Older Children (PAQ-C)